CLINICAL TRIAL: NCT02031978
Title: Women, Infant, and Children (WIC) Infant-Toddler Feeding Practices Study - II (ITFPS-2)
Brief Title: Feeding My Baby - A National WIC Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: USDA Food and Nutrition Service (U.S. Federal Agency)
Collaborators: Westat (Other); University of California, Los Angeles (Other); University of California, Berkeley (Other)
Responsible Party: Sponsor
Other Study IDs: AG3198B110020 & 12319820F006
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Breast Feeding; Infant Nutrition; Childhood Obesity; Infant Feeding Patterns; Feeding Behavior; Healthy Eating Index
Keywords: Breast Feeding; Infant Nutrition; Childhood Obesity; Infant feeding patterns; WIC; Diet quality; Food security
MeSH Terms: conditions — Breast Feeding; Pediatric Obesity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- WIC Program Participants: The cohort is made up of infants. Pregnant women enrolling in WIC for the first time for that pregnancy and mothers/caregivers of infants younger than 2.5 months of age enrolling in WIC for the first time are recruited to participate.

SUMMARY:
The goal of the study is to be a current examination of infant and toddler feeding practices among families receiving WIC services. It has been more than 10 years since the last study of such feeding practices, and in the interim important changes have taken place in the WIC program, in society, and in the science of nutrition. The study will include exploration of breastfeeding practices and support, more general feeding practices, nutritional intake of infants and toddlers, transitions in infant and toddler feeding practices, early precursors of obesity, and family factors that may influence all of these nutrition-related issues. It will also explore characteristics of the WIC program in selected sites, and how these relate to infant and toddler feeding decisions and practices. This study is important both to update knowledge about the WIC population, and to uncover possible new avenues of inquiry regarding early childhood obesity.

Update on November 25, 2020:

The WIC ITFPS-2 will now follow participants through child age 9 years. This unprecedented opportunity will provide FNS with a better understanding of the impact of WIC participation on health and nutrition outcomes in childhood.

DETAILED DESCRIPTION:
This observational study will employ a national probability sample of WIC participants and a longitudinal design to examine infant and toddler feeding behaviors and associated decision making. We will recruit and follow a core sample of infants and toddlers from birth through their second birthday and will oversample a supplemental group of WIC participants with low prevalence characteristics in the population to ensure representation of those groups (for instance, African-American mothers who breastfeed - a group with generally low levels of breastfeeding). The study will also gather information from key WIC Staff about the program, particularly about their breastfeeding policies and nutrition education activities. There are two categories of people from/about whom we will collect data - WIC Participants and WIC Program Representatives:

* WIC Participants: The target study participant is the infant/toddler, but we will recruit and conduct interviews with the mother (or primary caregiver), who are henceforth referred to as the participants. Participants must be at least 16 years old and parental consent and adolescent assent will be obtained for those under the age of majority in their state. The study will collect data about WIC participants in two ways:
* Interviews: Sampled WIC participants will be recruited and assigned to either a core or supplemental group. We will interview the core group up to thirteen times over a three-year period, with a prenatal interview (for those enrolled prenatally) and interviews every two months from the child's birth through age one, and about every three months between ages 1 and 2, and every 6 months between ages 2 and 3 (at ages 1, 3, 5, 7, 9, 11, 13, 15, 18, 24, 30 and 36 months). The supplemental group will only participate in four interviews (at ages 1 or 3, 7, 13, and 24 months). Study participants will also be asked at each interview about their child's food intake in the previous 24 hours using the USDA Automated Multiple Pass Method (AMPM) and supporting materials; and a 10 percent subsample of the core group will be asked to report a second day of intake 7-10 days after the initial interviews at 13, 15, 18, 24 and 36 months. The interviews will be conducted over the phone using a Computer-Assisted Telephone Interview (CATI).
* Health Data: The study will also collect data from hospital birth records on the infants' weight at birth; and from WIC administrative records on the infants' length and weight and WIC package prescription at four times during the study (at ages 6, 12, 24 and 36 months). When participants consent to enroll in the study, we will ask them to sign a Health Insurance Portability and Accountability Act (HIPAA) form releasing the records for the study. If a child in the core sample has dropped out of WIC, we will request data from their health care provider or ask the participant to travel to the nearest WIC site to be measured.
* WIC Program Representatives: Following the Sampling Plan described below the research team will recruit 80 WIC sites in 27 State Agencies to participate in the study and speak with them about the program.
* State and Local WIC Administrators: The study will conduct one, hour-long, semi-structured key informant interview with a State WIC administrator in each sampled State Agency, and a local WIC administrator for each sampled WIC site.
* WIC Site Staff: The study will also gather information from all staff (not to exceed 10) at sampled WIC sites through a one-time, 30-minute web-based survey.

The WIC enrollees will be sampled from a stratified, nationally representative sample of 80 WIC sites in 27 State Agencies. In addition to facilitating access to and creating efficient sampling frames for recruiting WIC participants, WIC program representatives in the WIC State and Local Agencies will provide important information to the study.

The study will use sampling methods to select the WIC site sample and the WIC participant sample. We will sample the lowest WIC unit that delivers services to WIC participants, called a "service site". Within each service site we will sample new WIC enrollees within a pre-determined recruitment window.

* Sampling WIC Service Sites. We plan a two-stage sampling approach that uses the WIC 2010 Participant Characteristics data (WIC PC 2010) to develop the WIC site sampling frame and a stratified sample design to select the sample of sites. In the first-stage we will use a group of characteristics to stratify the WIC sites into 40 strata. Because of uncertainties about the eligibility of the first-stage sampling units, these units will be selected in two phases. In the first phase a total of 160 sampling units in 42 State Agencies will be selected-4 from each of the 40 strata. After the phase 1 selection, we will list the service sites associated with each first-stage sampling unit selected and determine the eligibility of each unit. To be eligible for the study, a site must have an average minimum daily flow of 1.5 new WIC ITFPS-eligible enrollees per day and must be expected to remain in operation and enrolling new WIC participants during the WIC ITFPS recruitment period. In the second phase we will subsample eligible first-stage sampling units to arrive at the final sample of 80 first-stage sampling units (2 from each of the 40 strata). In first-stage sampling units that are local agencies with more than one eligible service site, a second stage of sampling will be conducted to select one service site. The final sample will consist of 80 eligible service sites. Once the second-stage sampling is complete, recruitment efforts will begin in earnest. Although due diligence will be used to recruit service sites, we anticipate that some sites may be unable or unwilling to cooperate. Such service sites will be replaced by members of a matched sample. This replacement of service sites by matched substitutes is similar to imputation.
* Sampling WIC participants within a sampled recruiting window. The WIC participant sample will be designed such that the total target number of sampled WIC enrollee is spread uniformly across the 80 sampled sites; that is, the recruitment of study participants will be designed so that each site will be expected to yield 98 sampled WIC enrollees. An important part of our sampling plan is the concept of recruiting "windows." A recruiting window will be a string of consecutive workdays during which we will be recruiting new WIC enrollees at each sampled service site. These windows will vary in length from 7 to 66 workdays. The length of the window will be pre-determined, based on typical daily enrollment volumes (obtained from the State following selection of the phase 1 sample of first-stage sampling units) and will be calculated in such a way as to yield an average of 98 sampled WIC enrollees per site. The 80 windows will be randomly assigned to a spread of starting dates across the 20-week field period for recruiting, with the pool of possible starting dates for a given site determined based on its average daily enrollments and enrollment schedule. Due to the variations in actual WIC enrollments over time, the actual number of sampled enrollees who enroll in WIC during the specified recruiting window will vary from site to site.

The full OMB package is available for review by visiting the Office of Management and Budget site at:

http://www.reginfo.gov/public/do/PRAViewICR?ref_nbr=201306-0584-008

OMB Control Number: 0584-0580

Update on November 25, 2020:

This observational study has been extended and will now follow children through age 9 years to examine the associations between prior WIC participation and children's health and nutrition outcomes. The core sample of participants will be interviewed 1, 3, 5, 7, 9, 11, 13, 15, 18, 24, 30, 36, 42, 48, 54, 60, and 72 months, and the supplemental sample will be interviewed at 1 or 3, 7, 13, 24, 30, 36, 42, 48, 54, 60, and 72 months; both core and supplemental sample participants will also receive a follow-up interview around the child's ninth birthday. In addition to the interviews at the aforementioned months, the study team will also ask participants to provide height and weight data around ages 6, 12, 24, 36, 48, 60, and 72 months and around age 9 years.

To date, all approved OMB information collection requests and associated documentation can be found at: https://www.reginfo.gov/public/Forward?SearchTarget=PRA&textfield=wic+infant+and+toddler+feeding+practices+study&Image61.x=24&Image61.y=11

ELIGIBILITY:
Inclusion Criteria:

* Enrolling in WIC for the first time for that pregnancy or infant
* Able to complete interviews in either English or Spanish

Exclusion Criteria:

* Having enrolled in WIC previously for that pregnancy or child
* The child being older than 2.5 months old at the time of recruitment
* Adolescent mothers under age 16 were not eligible to participate.\
* Adolescents who were in foster care at the time of enrollment were not eligible to participate, as foster parents cannot typically provide consent for research participation.
* Foster parents who were enrolling foster infants in WIC also were not eligible, as they cannot provide consent for the child's records.
* As defined by HHS regulations at 45 CFR part 46.303(c), prisoners were excluded from this research.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The target study participant is the infant. Mothers will be recruited prenatally and mothers/primary caregivers of infants will be recruited postnatally at 80 WIC clinic service locations.
Sampling Method: Probability Sample
Enrollment: 4367 (Actual)
Dates: Start 2013-07; Primary Completion 2023-07 (Estimated); Study Completion 2024-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Paolicelli, DrPH, Study Director — USDA Food and Nutrition Service; Christine Borger, PhD, Principal Investigator — Westat; Amanda Reat, PhD, Study Director — USDA Food and Nutrition Service

REFERENCES:
- [Result] Au LE, Gurzo K, Paolicelli C, Whaley SE, Weinfield NS, Ritchie LD. Diet Quality of US Infants and Toddlers 7-24 Months Old in the WIC Infant and Toddler Feeding Practices Study-2. J Nutr. 2018 Nov 1;148(11):1786-1793. doi: 10.1093/jn/nxy192. PMID 30383276
- [Result] Au LE, Paolicelli C, Gurzo K, Ritchie LD, Weinfield NS, Plank KR, Whaley SE. Contribution of WIC-Eligible Foods to the Overall Diet of 13- and 24-Month-Old Toddlers in the WIC Infant and Toddler Feeding Practices Study-2. J Acad Nutr Diet. 2019 Mar;119(3):435-448. doi: 10.1016/j.jand.2018.11.001. Epub 2019 Jan 9. PMID 30638822
- [Result] Whaley SE, Martinez CE, Paolicelli C, Ritchie LD, Weinfield NS. Predictors of WIC Participation Through 2 Years of Age. J Nutr Educ Behav. 2020 Jul;52(7):672-679. doi: 10.1016/j.jneb.2019.12.015. Epub 2020 Feb 14. PMID 32067886
- [Result] Gleason S, Wilkin MK, Sallack L, Whaley SE, Martinez C, Paolicelli C. Breastfeeding Duration Is Associated With WIC Site-Level Breastfeeding Support Practices. J Nutr Educ Behav. 2020 Jul;52(7):680-687. doi: 10.1016/j.jneb.2020.01.014. Epub 2020 Mar 11. PMID 32171671
- [Result] Weinfield NS, Borger C, Gola AA. Breastfeeding Duration in a Low-Income Sample Is Associated With Child Diet Quality at Age Three. J Hum Lact. 2021 Feb;37(1):183-193. doi: 10.1177/0890334420903029. Epub 2020 Feb 24. PMID 32091965
- [Result] Weinfield NS, Borger C, Au LE, Whaley SE, Berman D, Ritchie LD. Longer Participation in WIC Is Associated with Better Diet Quality in 24-Month-Old Children. J Acad Nutr Diet. 2020 Jun;120(6):963-971. doi: 10.1016/j.jand.2019.12.012. Epub 2020 Feb 14. PMID 32067936
- [Result] Hamner HC, Beauregard JL, Li R, Nelson JM, Perrine CG. Meeting breastfeeding intentions differ by race/ethnicity, Infant and Toddler Feeding Practices Study-2. Matern Child Nutr. 2021 Apr;17(2):e13093. doi: 10.1111/mcn.13093. Epub 2020 Oct 1. PMID 33006242
- [Result] Anderson CE, Martinez CE, Ventura AK, Whaley SE. Potential overfeeding among formula fed Special Supplemental Nutrition Program for Women, Infants and Children participants and associated factors. Pediatr Obes. 2020 Dec;15(12):e12687. doi: 10.1111/ijpo.12687. Epub 2020 Jun 18. PMID 32558255
- [Result] Borger C, Paolicelli C, Ritchie L, Whaley SE, DeMatteis J, Sun B, Zimmerman TP, Reat A, Dixit-Joshi S. Shifts in Sources of Food but Stable Nutritional Outcomes among Children in the Early Months of the COVID-19 Pandemic. Int J Environ Res Public Health. 2021 Nov 30;18(23):12626. doi: 10.3390/ijerph182312626. PMID 34886351
- [Result] Weinfield NS, Anderson CE. Postpartum Symptoms of Depression are Related to Infant Feeding Practices in a National WIC Sample. J Nutr Educ Behav. 2022 Feb;54(2):118-124. doi: 10.1016/j.jneb.2021.09.002. Epub 2021 Dec 18. PMID 34930709
- [Result] Thompson HR, Borger C, Paolicelli C, Whaley SE, Reat A, Ritchie L. The Relationship between Breastfeeding and Initial Vegetable Introduction with Vegetable Consumption in a National Cohort of Children Ages 1-5 Years from Low-Income Households. Nutrients. 2022 Apr 22;14(9):1740. doi: 10.3390/nu14091740. PMID 35565708
- [Result] Borger C, Paolicelli CP, Sun B. Duration of Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) Participation is Associated With Children's Diet Quality at Age 3 Years. Am J Prev Med. 2022 Jun;62(6):e343-e350. doi: 10.1016/j.amepre.2021.12.019. Epub 2022 Mar 8. PMID 35277313
- [Result] Bably MB, Paul R, Laditka SB, Racine EF. Factors Associated with the Initiation of Added Sugar among Low-Income Young Children Participating in the Special Supplemental Nutrition Program for Women, Infants, and Children in the US. Nutrients. 2021 Oct 29;13(11):3888. doi: 10.3390/nu13113888. PMID 34836143
- [Result] Chaparro MP, Anderson CE. Differences in Early Childhood Dietary Behaviors by Infant Feeding Type and Sex. J Nutr. 2021 Jul 1;151(7):2001-2009. doi: 10.1093/jn/nxab076. PMID 33847341
- [Result] Bably MB, Laditka SB, Paul R, Racine EF. Age of Bottle Cessation and BMI-for-Age Percentile among Children Aged Thirty-Six Months Participating in WIC. Child Obes. 2022 Apr;18(3):197-205. doi: 10.1089/chi.2021.0119. Epub 2021 Sep 22. PMID 34551266
- [Result] Beauregard JL, Nelson JM, Li R, Perrine CG, Hamner HC. Maternity Care Practices and Breastfeeding Intentions at One Month Among Low-Income Women. Pediatrics. 2022 Apr 1;149(4):e2021052561. doi: 10.1542/peds.2021-052561. PMID 35253063
- [Result] Hamner HC, Chiang KV, Li R. Returning to Work and Breastfeeding Duration at 12 Months, WIC Infant and Toddler Feeding Practices Study-2. Breastfeed Med. 2021 Dec;16(12):956-964. doi: 10.1089/bfm.2021.0081. Epub 2021 Jul 28. PMID 34319808
- [Result] Thompson IJB, Ritchie LD, Bradshaw PT, Mujahid MS, Au LE. Earlier Introduction to Sugar-Sweetened Beverages Associated With Lower Diet Quality Among WIC Children at Age 3 Years. J Nutr Educ Behav. 2021 Nov;53(11):912-920. doi: 10.1016/j.jneb.2021.04.468. Epub 2021 Jul 3. PMID 34229969
- [Result] Paolicelli C, Berman D, Owens T, Magness A, Scanlon KS. Breastfeeding and Complementary Feeding Patterns Among Women Enrolled in WIC: WIC Infant and Toddler Feeding Practices Study-2. Breastfeed Med. 2017 Oct;12(8):482-486. doi: 10.1089/bfm.2017.0118. Epub 2017 Aug 22. No abstract available. PMID 28829156
- [Derived] Chaney AM, Arnold CD, Frongillo EA, Ritchie LD, Steele EM, Au LE. Infant diet quality index predicts nutrients of concern and ultra-processed food intake in low-income children in the United States. Curr Dev Nutr. 2024 Oct 18;8(11):104483. doi: 10.1016/j.cdnut.2024.104483. eCollection 2024 Nov. PMID 39610764
- [Derived] Borger C, Weinfield NS, Paolicelli C, Sun B, May L. Prenatal and Postnatal Experiences Predict Breastfeeding Patterns in the WIC Infant and Toddler Feeding Practices Study-2. Breastfeed Med. 2021 Nov;16(11):869-877. doi: 10.1089/bfm.2021.0054. Epub 2021 Jul 15. PMID 34265220
- [Derived] Harrison GG, Hirschman JD, Owens TA, McNutt SW, Sallack LE. WIC Infant and Toddler Feeding Practices Study: protocol design and implementation. Am J Clin Nutr. 2014 Mar;99(3):742S-6S. doi: 10.3945/ajcn.113.073585. Epub 2014 Jan 29. PMID 24477040
- See also: WIC ITFPS-2: Intentions to Breastfeed Report — https://www.fns.usda.gov/wic/special-supplemental-nutrition-program-women-infants-and-children-wic-infant-and-toddler-feeding
- See also: WIC ITFPS-2: Infant Year Report — https://www.fns.usda.gov/wic/wic-infant-and-toddler-feeding-practices-study-2-infant-year-report
- See also: WIC ITFPS-2: Second Year Report — https://www.fns.usda.gov/wic/wic-infant-and-toddler-feeding-practices-study-2-second-year-report
- See also: WIC ITFPS-2: Third Year Report — https://www.fns.usda.gov/wic/wic-infant-and-toddler-feeding-practices-study-2-third-year-report
- See also: WIC ITFPS-2: Fourth Year Report — https://www.fns.usda.gov/wic/infant-and-toddler-feeding-practices-study-2-fourth-year-report

RESULTS

PARTICIPANT FLOW:
Groups:
- WIC Participants: Mothers and their child (mother-child dyads)
Period: Overall Study
Arm/Group | WIC Participants
Started | 4367
Completed | 4367
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The Main Analysis sample includes 3,777 cases that have completed a 1- and/or 3-month interview.
Arm/Group | WIC Participants
Number analyzed (Participants) | 4367
Age, Customized [Count of Participants; unit: Participants] — Age of study child's mother at baseline
  Participants
    Age of Mother: 16-19y | 446
    Age of Mother: 20-25y | 1569
    Age of Mother: 26y+ | 1762
    Age of Mother: Missing | 590
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of the study child at birth Population: Missing/unknown = 356 participants
  Participants
    number analyzed (Participants) | 4011
    Female | 2054
    Male | 1957
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1443
  Not Hispanic or Latino | 2,329
  Unknown or Not Reported | 595

OUTCOME MEASURES:

1. Primary Outcome: Breastfeeding Initiation
Description: Whether the mother initiated breastfeeding after child was born
Time Frame: first month after birth of child
Measure: Count of Participants; unit: Participants
Arm/Group | WIC Participants
Number analyzed (Participants) | 3777
Participants
  Mothers who did initiate breastfeeding | 3152
  Mothers who did not initiate breastfeeding | 625

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | WIC Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2012-09-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT02031978/Prot_SAP_000.pdf
  • Informed Consent Form (2014-06-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT02031978/ICF_001.pdf